CLINICAL TRIAL: NCT01128036
Title: Comparison of Different Locations for Pulse Oximetry Probes in Adult Cardiovascular Patients With Poor Peripheral Perfusion
Brief Title: Comparison of Different Locations for Pulse Oximetry Probes in Cardiovascular (CV) Patients With Poor Peripheral Perfusion
Status: Terminated | Type: Observational
Why Stopped: Terminated due to software issues.
Sponsor: Saint Luke's Health System (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Marci Sportsman, Saint Luke's Hospital
Other Study IDs: COVMOPO0054
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Congestive Heart Failure; Cardiomyopathy
Keywords: Congestive Heart failure; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHF, cardomyopathy: Patients with signs of poor peripheral perfusion due to cardiomyopathy or congestive heart failure

SUMMARY:
The purpose of this study is to determine if the forehand location for sensor placement has less episodes of signal dropout than the finger sensor location. In addition, this study will evaluate two finger sensors, which utilize different technology to compare signal quality.

DETAILED DESCRIPTION:
A comparison study design will be used to evaluate the signal quality of pulse oximetry sensors placed in two locations: forehand and finger. Each subject will serve as their own control, with measurements of signal quality evaluated at 2 second intervals over a period of one hour. The measurements will be recorded simultaneously with a computer program and laptop computer. Finger and forehand sensors will be applied according to manufacturer's guidelines. An output connection will be made from each pulse oximeter computer unit to a password protected, laptop computer for data downloading. Data will be collected for a 1 hour period at 2 second increments and stored in the hard drive of the laptop. Following completion of data collection, the study sensors will be removed.

ELIGIBILITY:
Inclusion Criteria:

* CICU patients with a new diagnosis or history of CHF or cardiomyopathy
* Patients with a medical order for pulse oximetry monitoring
* Age greater than or equal to 18 years of age
* English speaking
* Signs of hypoperfusion

Exclusion Criteria:

* CICU patients with an impediment to sensor application
* CICU patients with excessive facial edema
* CICU patients with mechanical ventilation
* CICU patients with intra-aortic balloon pump therapy
* CICU patients with intravenous vasopressor drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the CICU (Coronary Intensive Coronary Unit) with congestive heart failure or cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Signal quality loss (dropout rate) | Every 2 seconds for one hour

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Riggs, MSN, Study Director — Saint Luke's Hospital; Marci Sportsman, BSN, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital, Kansas City, Missouri, United States